CLINICAL TRIAL: NCT04983056
Title: Fournier's Gangrene: Seven Years of Experience in the Emergencies Service of Visceral Surgery at Ibn Rochd UHC
Brief Title: Management of Fournier Gangrene at Ibn Rochd University Hospital Center
Status: Completed | Type: Observational
Sponsor: Sylvestre KABURA (Other)
Responsible Party: Sponsor-Investigator, Sylvestre KABURA, Principal investigator, Centre Hospitalier Universitaire Ibn Rochd
Organization: Centre Hospitalier Universitaire Ibn Rochd (Other)
Other Study IDs: FZBKSMP35
Record Dates: First submitted 2021-07-07; First posted 2021-07-30 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Fournier Gangrene
Keywords: Fournier's Gangrene, stoma, necrosectomy
MeSH Terms: conditions — Fournier Gangrene

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: None Retained — The pus from purulent and necrotized tissues

INTERVENTIONS:
Procedure: Necrotesectomy associated with cleanleness stoma — Excision of all necrotised tissues after stool diversion and wound dressing using

SUMMARY:
Case series with retrospective data collection of patients treated for Fournier's gangrene between January 2010 and March 2017. The main etiologies, risk factors, postoperative complications outcomes and long term follow up results were analyzed.

DETAILED DESCRIPTION:
Eight four (84) patients were recruited. The average age of our patients was 49 years (with limits of 20 to 76), the male gender dominates our series (83.33%) with a sex ratio of 5M / 1W, the most frequently found risk factor was diabetes mellitus (37%). The most common etiology was anal abscesses (32%). The average time to consultation was 8 days (limits ranges from 3 to 30 days). All patients were admitted at a necrosis stage (100%). Anemia was identified in 85% of cases. The low platelets were noticed in 44.03% of cases. Hypoalbuminemia was found in 93% of cases. All patients (100%) benefited resuscitation initially and antibiotic therapy on their admission. They received emergency surgical debridement with a cleansing stoma. The average length of hospital stay was 13 days and complications occurred in 33% of cases. The mortality rate was 7.14%. then we conclude that Fournier's gangrene is a medico-surgical emergency with a high morbidity and mortality rate. Early diagnosis as well as antibiotic therapy and the quality of debridement save the patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Fournier Gangrene

Exclusion Criteria:

* Other perineal diseases which are differential diagnosis of Fournier gangrene

Ages: 15 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: . Patients with Fournier Gangrene
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2021-07-02 (Actual)

PRIMARY OUTCOMES:
Number of patients who died for fournier gangrene | Six months
  The mortality rate of patients with Fournier Gangrene after six months

IPD SHARING:
Plan to Share IPD: Undecided